CLINICAL TRIAL: NCT04154358
Title: Implementing HPV DNA Self-Collection to Increase Rates of Cervical Cancer Screening in Transgender Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augusta University (Other)
Collaborators: The Equality Clinic of Augusta (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1410051-2
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Transgenderism; Cervical Cancer; Human Papilloma Virus
MeSH Terms: conditions — Transsexualism; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HPV Testing (Experimental): Will perform HPV testing with self-collected specimen
  Interventions: Diagnostic Test: HPV testing

INTERVENTIONS:
Diagnostic Test: HPV testing — will perform HPV testing with self-collected specimen

SUMMARY:
Transgender men are individuals born genetically female that have a gender identity that is incongruent with their biological sex. For those who have begun or completed transition, they may present as males but still have a uterus and cervix. Thus far, no distinction has been made between routine cervical cancer screening guidelines in non-transgender women and those for transgender men, despite wide variations in sexual practices, including lifelong vaginal abstinence. The purpose of this study is to offer transgender men seen at clinic visits self-collected HPV testing to evaluate for improved cervical cancer screening rates, as well as a survey to further investigate sexual practices, rates of appropriate screening prior to being offered self-collection, and barriers to obtaining appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 for survey and age> 25 for HPV testing
* Transgender male or gender non-conforming identity
* Female sex at birth
* Consent to participate in the study

Exclusion Criteria:

* impaired decision making capacity
* Absence of cervix
* Non-English speaking

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be transgender masculine identifying with uterus and cervix.
Enrollment: 100 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of cervical cancer screening | 1 year
  Evaluate whether implementation of HPV DNA self swabs will increase rates of cervical cancer screening among transgender men by percentage of trans men who obtain screening through the study

SECONDARY OUTCOMES:
incidence of barriers to care | 1 year
  Determine which barriers contribute most to lack of cervical cancer screening among transgender men. Measured via survey.
incidence of high risk sexual practices | 1 year
  Evaluate for the presence of high risk behaviors to determine whether transgender men in our population are at higher or lower risk for HPV-related cervical dysplasia. Measured via survey.
rate of HPV vaccination | 1 year
  Evaluate percentage of transgender men that have been vaccinated for HPV. Measured via survey.

IPD SHARING:
Plan to Share IPD: No